CLINICAL TRIAL: NCT01090024
Title: A Randomised, Double-blind, Placebo-controlled, Efficacy and Safety Cross-over Study of 4 Weeks of Oral BI 671800 ED 200 mg Twice Daily or 400 mg Once Daily Administered in the Morning (AM) or Evening (PM), in Symptomatic Asthma Patients on Inhaled Fluticasone Propionate MDI
Brief Title: Bi 671800 in Asthmatic Patients on Inhaled Corticosteroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1268.53
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — BI 671800

ARMS (4):
- BI 671800 AM and PM (Experimental): Patients receiving two capsules twice daily
  Interventions: Drug: BI 671800
- BI 671800 AM (Experimental): Patients receiving four capsules in the morning
  Interventions: Drug: BI 671800
- BI 671800 PM (Experimental): Patients receiving four capsules in the evening
  Interventions: Drug: BI 671800
- Placebo (Placebo Comparator): Patients receiving four capsules twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 671800 — BI 671800
  Arms: BI 671800 AM; BI 671800 AM and PM; BI 671800 PM
Drug: Placebo — Placebo matching BI 671800
  Arms: Placebo

SUMMARY:
To investigate the effectiveness and safety of BI 671800 given in the morning (AM), evening (PM) or twice daily (b.i.d.) compared too placebo as add on therapy to inhaled corticosteroid in symptomatic asthma patients.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent consistent with International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP) (ICH-GCP)
2. Three month history of reversible (12% with 200 mL) asthma according to [Global Initiative for Asthma (GINA)] with following spirometry at randomization:forced expiratory volume in 1 second (FEV1) 60%-85%.
3. Stable inhaled corticosteroid (ICS) dose 3 months prior to screening.
4. Diagnosis of asthma prior to 40 years.
5. Asthma Control Questionnaire (ACQ) at least 1.5 at randomization.
6. Male or female, 18 to 65 years.
7. Non-smokers or ex-smokers ( less than 10 pack year history) with negative cotinine screen.
8. Able to perform pulmonary function test (PFT).

Exclusion criteria:

1. Significant diseases other than asthma or allergic rhinitis.
2. Hepatic transaminases or total bilirubin greater than 1.5 upper limit of normal (ULN).
3. Hospitalizations for asthma or asthma related intubation within 3 months.
4. Uncontrolled asthma on ICS + another controller.
5. Respiratory tract infection or exacerbation within 4 weeks.
6. FEV1 less than 40%, more than 12 puffs of short acting beta agonists (SABA) on more than two consecutive days or asthma exacerbation during the run-in period.
7. Participation in another interventional study.
8. Pregnant or nursing women.
9. Women of child bearing potential nor using appropriate methods of birth control as defined by protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2011-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (14):
- United States (14):
  - 1268.53.01013 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1268.53.01014 Boehringer Ingelheim Investigational Site, Mission Viejo, California
  - 1268.53.01002 Boehringer Ingelheim Investigational Site, Stockton, California
  - 1268.53.01009 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1268.53.01011 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1268.53.01001 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1268.53.01005 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1268.53.01006 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1268.53.01007 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1268.53.01010 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1268.53.01003 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1268.53.01008 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 1268.53.01012 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1268.53.01015 Boehringer Ingelheim Investigational Site, Richmond, Virginia

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomised, double-blind, placebo-controlled, cross-over study was to investigate efficacy and safety of 3×4-week treatment periods of oral BI 671800 Ethylenediamine 200 milligram (mg) twice or 400 mg once daily administered in the morning or evening, in symptomatic asthma patients on inhaled fluticasone propionate Metered Dose Inhaler.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 400mg PM QD (C): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks.
- Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 200 mg BID (D): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks.
- Placebo(A)/BI 671800 400mg PM QD (C)/BI 671800 400mg AM QD (B): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks.
- Placebo (A)/BI 671800 400mg PM QD (C)/BI 671800 200 mg BID (D): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks.
- Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks.
- Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks.
- BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 400 mg PM QD(C): (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks.
- BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 200 mg BID(D): (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks.
- BI 671800 400 mg AM QD(B)/BI 671800 400 mg PM QD(C)/Placebo(A): (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
- BI 671800 400 mg AM QD(B)/BI 671800 200 mg BID(D)/Placebo(A): (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
- BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 400 mg AM QD(B): (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks.
- BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 200 mg BID(D): (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks.
- BI 671800 400 mg PM QD(C)/BI 671800 400 mg AM QD(B)/Placebo(A): (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
- BI 671800 400 mg PM QD(C)/BI 671800 200 mg BID(D)/Placebo(A): (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
- BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg AM QD(B): (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks.
- BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg PM QD(C): (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks.
- BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B)/Placebo(A): (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
- BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C)/Placebo(A): (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks, followed by (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks, followed by (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
Period: Period 1
Arm/Group | Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 400mg PM QD (C) | Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 200 mg BID (D) | Placebo(A)/BI 671800 400mg PM QD (C)/BI 671800 400mg AM QD (B) | Placebo (A)/BI 671800 400mg PM QD (C)/BI 671800 200 mg BID (D) | Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B) | Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C) | BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 400 mg PM QD(C) | BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 200 mg BID(D) | BI 671800 400 mg AM QD(B)/BI 671800 400 mg PM QD(C)/Placebo(A) | BI 671800 400 mg AM QD(B)/BI 671800 200 mg BID(D)/Placebo(A) | BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 400 mg AM QD(B) | BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 200 mg BID(D) | BI 671800 400 mg PM QD(C)/BI 671800 400 mg AM QD(B)/Placebo(A) | BI 671800 400 mg PM QD(C)/BI 671800 200 mg BID(D)/Placebo(A) | BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg AM QD(B) | BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg PM QD(C) | BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B)/Placebo(A) | BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C)/Placebo(A)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Met exclusion criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 400mg PM QD (C) | Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 200 mg BID (D) | Placebo(A)/BI 671800 400mg PM QD (C)/BI 671800 400mg AM QD (B) | Placebo (A)/BI 671800 400mg PM QD (C)/BI 671800 200 mg BID (D) | Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B) | Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C) | BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 400 mg PM QD(C) | BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 200 mg BID(D) | BI 671800 400 mg AM QD(B)/BI 671800 400 mg PM QD(C)/Placebo(A) | BI 671800 400 mg AM QD(B)/BI 671800 200 mg BID(D)/Placebo(A) | BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 400 mg AM QD(B) | BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 200 mg BID(D) | BI 671800 400 mg PM QD(C)/BI 671800 400 mg AM QD(B)/Placebo(A) | BI 671800 400 mg PM QD(C)/BI 671800 200 mg BID(D)/Placebo(A) | BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg AM QD(B) | BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg PM QD(C) | BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B)/Placebo(A) | BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C)/Placebo(A)
Started | 6 | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
Completed | 5 | 5 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 400mg PM QD (C) | Placebo(A)/BI 671800 400mg AM QD (B)/BI 671800 200 mg BID (D) | Placebo(A)/BI 671800 400mg PM QD (C)/BI 671800 400mg AM QD (B) | Placebo (A)/BI 671800 400mg PM QD (C)/BI 671800 200 mg BID (D) | Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B) | Placebo(A)/BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C) | BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 400 mg PM QD(C) | BI 671800 400 mg AM QD(B)/Placebo(A)/BI 671800 200 mg BID(D) | BI 671800 400 mg AM QD(B)/BI 671800 400 mg PM QD(C)/Placebo(A) | BI 671800 400 mg AM QD(B)/BI 671800 200 mg BID(D)/Placebo(A) | BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 400 mg AM QD(B) | BI 671800 400 mg PM QD(C)/Placebo(A)/BI 671800 200 mg BID(D) | BI 671800 400 mg PM QD(C)/BI 671800 400 mg AM QD(B)/Placebo(A) | BI 671800 400 mg PM QD(C)/BI 671800 200 mg BID(D)/Placebo(A) | BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg AM QD(B) | BI 671800 200 mg BID(D)/Placebo(A)/BI 671800 400 mg PM QD(C) | BI 671800 200 mg BID(D)/BI 671800 400 mg AM QD(B)/Placebo(A) | BI 671800 200 mg BID(D)/BI 671800 400 mg PM QD(C)/Placebo(A)
Started | 5 | 5 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
Treated | 5 | 5 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 5 | 5 | 6 | 5
Completed | 5 | 5 | 6 | 4 | 6 | 5 | 6 | 6 | 5 | 5 | 6 | 5 | 6 | 6 | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All patients treated with at least one dose of blinded study drug.
Groups:
- Overall Population: All of the enrolled participants that were randomized to one of the treatment sequences for 3 × 4-week treatment periods and treated with at least one dose of study drug.
Arm/Group | Overall Population
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 89
  More than one race | 0
  Unknown or Not Reported | 0
Trough forced expiratory volume in one second (FEV1) percent predicted [Mean (Standard Deviation); unit: Percentage of predicted trough FEV1] — Baseline trough FEV1 percent (%) predicted was defined as the mean of FEV1 % predicted trough values taken at 25 minutes and 10 minutes prior to the first dose of randomized treatment. Population: Treated set: All patients treated with at least one dose of blinded study drug. Participants in treated set with non-missing baseline (Week 0) trough FEV1 percent predicted values were included.
  Percentage of predicted trough FEV1
    number analyzed (Participants) | 107
    (all) | 72.816 (7.5759)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Trough Forced Expiratory Volume in One Second (FEV1) Percent Predicted After 4 Weeks of Treatment
Description: Trough FEV1 percent (%) predicted was defined as the mean of the morning and the evening FEV1 % predicted daily trough value at the end of the dosing interval. For the morning (evening) measurements, when FEV1 % predicted was available at both 25 minutes and 10 minutes prior to morning (evening) test-drug inhalation, morning (evening) trough FEV1 % predicted was the mean of these two morning (evening) pre-inhalation measurements. Trough FEV1 % predicted change from baseline after 4 weeks of treatment was defined as the change from baseline in the mean of the morning and the evening trough FEV1 % predicted.
Time Frame: At baseline and 4 weeks
Population: Full analysis set (FAS): All patients randomized, treated with at least one dose of blinded study drug, with a baseline Forced expiratory volume in one second (FEV1) value and at least one on-treatment trough FEV1 value. The FAS is the basis for the intention-to-treat analysis. Participants with non-missing endpoint measurements were included.
Measure: Mean (Standard Error); unit: Percentage of predicted trough FEV1
Groups:
- Placebo (A): (A) 4 capsules of 100 milligram (mg) of BI 671800 Ethylenediamine (ED) matching placebo (Total 400 mg) administered orally once daily in the morning or 4 capsules of 100 milligram (mg) of BI 671800 ED matching placebo (Total 400 mg) administered orally once daily in the evening for a treatment period of 4 weeks.
- BI 671800 400mg AM QD (B): (B) 4 capsules of 100 milligram (mg) BI 671800 Ethylenediamine (ED) (Total 400 mg) were administered orally once daily (QD) in the morning (AM) for a treatment period of 4 weeks.
- BI 671800 400mg PM QD (C): (C) 4 capsules of 100 milligram (mg) BI 671800 ED (Total 400 mg) were administered orally once daily (QD) in the evening (PM) for a treatment period of 4 weeks.
- BI 671800 200mg BID (D): (D) 2 capsules of 100 milligram (mg) BI 671800 ED (Total 200 mg) were administered orally twice daily (BID) in the morning and in the evening for a treatment period of 4 weeks.
Arm/Group | Placebo (A) | BI 671800 400mg AM QD (B) | BI 671800 400mg PM QD (C) | BI 671800 200mg BID (D)
Number analyzed (Participants) | 100 | 68 | 64 | 64
Percentage of predicted trough FEV1 | 0.128 (0.536) | 0.409 (0.612) | 0.798 (0.626) | 0.211 (0.626)
Statistical Analysis 1: Comparison: Placebo (A) vs BI 671800 200mg BID (D); Restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM) with terms for baseline, treatment and period as fixed effects and patient as a random effect was used. A compound symmetry covariance structure was used; Test type: Superiority — One-sided p-value testing superiority of BI 671800 vs placebo with 2.5% alpha; p = 0.4473, Mixed effect model; Adjusted means difference = 0.083, 95% CI 2-sided [-1.147 to 1.313], Standard Error of Mean 0.624 — Adjusted means difference of BI 671800 200 mg BID (D) vs Placebo (A)
Statistical Analysis 2: Comparison: Placebo (A) vs BI 671800 400mg PM QD (C); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — One-sided p-value testing superiority of BI 671800 vs placebo with 2.5% alpha; p = 0.1426, Mixed effect model; Adjusted means difference = 0.670, 95% CI 2-sided [-0.563 to 1.903], Standard Error of Mean 0.625 — Adjusted means difference of BI 671800 400 mg PM QD (C) vs Placebo (A)
Statistical Analysis 3: Comparison: Placebo (A) vs BI 671800 400mg AM QD (B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority — One-sided p-value testing superiority of BI 671800 vs placebo with 2.5% alpha; p = 0.3231, Mixed effect model; Adjusted means difference = 0.281, 95% CI 2-sided [-0.924 to 1.486], Standard Error of Mean 0.611 — Adjusted means difference of BI 671800 400 mg AM QD (B) vs Placebo (A)

2. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Mean Score After Four Weeks of Treatment
Description: The Asthma Control Questionnaire (ACQ) consists of 6 patient self-evaluated questions and 1 by clinical staff with each question in 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of less than or equal to 0.75 indicate well-controlled asthma, scores between 0.76 and less than 1.5 indicate partly controlled asthma, and a score greater than or equal to 1.5 indicates uncontrolled asthma.
Time Frame: At baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (A) | BI 671800 400mg AM QD (B) | BI 671800 400mg PM QD (C) | BI 671800 200mg BID (D)
Number analyzed (Participants) | 101 | 68 | 64 | 64
Score on a scale | -0.595 (0.059) | -0.688 (0.066) | -0.621 (0.068) | -0.651 (0.068)
Statistical Analysis 1: Comparison: Placebo (A) vs BI 671800 200mg BID (D); Restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM) with terms for baseline, treatment and period as fixed effects and patient as a random effect was used. A autoregressive covariance structure was used; Test type: Superiority — One-sided p-value testing superiority of BI 671800 vs placebo with 2.5% alpha; p = 0.1879, Mixed effect model; Adjusted means difference = -0.056, 95% CI 2-sided [-0.180 to 0.068], Standard Error of Mean 0.063 — Adjusted means difference of BI 671800 200 mg BID (D) vs Placebo (A)
Statistical Analysis 2: Comparison: Placebo (A) vs BI 671800 400mg PM QD (C); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — One-sided p-value testing superiority of BI 671800 vs placebo with 2.5% alpha; p = 0.3384, Mixed effect model; Adjusted means difference = -0.026, 95% CI 2-sided [-0.151 to 0.098], Standard Error of Mean 0.063 — Adjusted means difference of BI 671800 400 mg PM QD (C) vs Placebo (A)
Statistical Analysis 3: Comparison: Placebo (A) vs BI 671800 400mg AM QD (B); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — One-sided p-value testing superiority of BI 671800 vs placebo with 2.5% alpha; p = 0.0670, Mixed effect model; Adjusted means difference = -0.093, 95% CI 2-sided [-0.214 to 0.029], Standard Error of Mean 0.062 — Adjusted means difference of BI 671800 400 mg AM QD (B) vs Placebo (A)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 4 weeks thereafter, up to 4 weeks + 5 days for (serious) adverse events, up to 4 weeks + 2 weeks of follow-up for all-cause mortality.
Description: Treated set: All patients treated with at least one dose of blinded study drug. Total number of participants per treatment is lower than the total started number of participants due to participants having left the sequence before being exposed to the respective treatment.
Arm/Group | Placebo (A) | BI 671800 400mg AM QD (B) | BI 671800 400mg PM QD (C) | BI 671800 200mg BID (D)
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/70 | 0/68 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/70 | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 4/104 | 3/70 | 5/68 | 2/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (A) (N=104) | BI 671800 400mg AM QD (B) (N=70) | BI 671800 400mg PM QD (C) (N=68) | BI 671800 200mg BID (D) (N=67)
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.